CLINICAL TRIAL: NCT01451931
Title: Randomized Controlled Trial of Ultrasound Versus CT (Computed Tomography) for Patients in the Emergency Department With Suspected Renal Colic
Brief Title: Study of Tomography of Nephrolithiasis Evaluation
Acronym: STONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RSB-1002670
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Urolithiasis
Keywords: kidney stone; urolithiasis; urinary tract infection; ultrasound; computed tomography; safety; cost; accuracy
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Point-of-care Ultrasound (Experimental): Patient with suspected urolithiasis will receive ultrasonography performed in the emergency department. Perform ultrasonography in the ED (physician).
  Interventions: Other: Point-of-care Ultrasound
- Radiology Ultrasound (Experimental): Patient with suspected urolithiasis will receive diagnostic ultrasonography in the radiology department. Diagnostic ultrasound completed in the radiology department at time 0.
  Interventions: Radiation: Radiology Ultrasound
- Radiology CT (Experimental): Patient with suspected urolithiasis will receive computed tomography in the radiology department. Computed tomography of abdomen completed in the radiology department at time 0.
  Interventions: Other: Radiology CT

INTERVENTIONS:
Other: Point-of-care Ultrasound — Perform ultrasonography in the ED (physician).
  Arms: Point-of-care Ultrasound
Radiation: Radiology Ultrasound — Diagnostic ultrasound completed in the radiology department at time 0.
  Arms: Radiology Ultrasound
Other: Radiology CT — Computed tomography of abdomen completed in the radiology department at time 0.
  Arms: Radiology CT

SUMMARY:
This is a multi-center, randomized controlled trial of ultrasonography (ultrasound) compared to computed tomography (CT) for the initial emergency room evaluation of patients with suspected renal colic. The investigators will compare several measures of effectiveness including morbidity related to the patient's underlying disease, or complications related to delayed diagnosis, patient status regarding pain/missed days of work, and utilization of health care resources based on one of three study arms: ultrasound in the Emergency Department, ultrasound in Radiology or CT.

DETAILED DESCRIPTION:
This is a multi-center, randomized controlled trial of ultrasonography compared with computed tomography (CT) for the evaluation of patients with suspected urolithiasis. The study will be conducted at 15 large urban Emergency Departments (EDs), reflecting geographic, socioeconomic, racial and ethnic diversity, and include academic medical centers as well as safety net hospitals. The patients will be randomized to one of three arms: 1) ultrasound in the Emergency Department (ED), 2) ultrasound in radiology or 3) CT in radiology. The investigators will then collect precise and unbiased data on a comprehensive range of outcomes that will allow assessment of effectiveness, safety, accuracy and cost between patients randomized to one the three groups. Taken together, these measures are intended to provide the basis for a valid comparison of imaging of patients with suspected urolithiasis seen in the ED. The results of this trial could lead to a change in clinical practice that is associated with both improved patient outcomes and reduced cost. Broad stakeholder involvement from within radiology, emergency medicine and several subspecialty communities has been sought to ensure the strategic completion of study aims and to help rapidly disseminate the results of the study into clinical practice. This will create a collaborative network of EDs willing to act as a laboratory for studying the comparative effectiveness of diagnostic testing. As a result, the proposed trial will demonstrate the feasibility of conducting Randomized Control Trials (RCTs) of imaging that incorporates measurements of outcomes that can be expanded to additional imaging tests in the future.

ELIGIBILITY:
Inclusion Criteria:

* men or women = or >18 but <76 years of age presenting with acute renal colic
* Emergency department physician highly suspects a primary diagnosis of kidney stones (renal colic) or the patient requires imaging to rule out kidney stones.

Exclusion Criteria:

* children < 18 years old
* elderly patients > or = 76 years old
* pregnancy or planning pregnancy
* Morbid obesity (>285 pounds in men, >250 pounds in women)
* patients with an acute abdomen, signs of sepsis, signs of alternate diagnosis (ie appendicitis, abdominal aortic aneurysm, pyelonephritis, kidney stones not suspected).
* history of kidney problems (hemodialysis, kidney transplant, presence of only one kidney)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2776 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Smith-Bindman, MD, Principal Investigator — University of California, San Francisco, Department of Radiology and Biomedical Imaging; Clifford Rosen, MD, Study Chair — Professor of Medicine, Tufts University (Data Safety Monitoring Board Chair)
Locations (15):
- United States (15):
  - UCSF at Fresno, Fresno, California
  - University of California, Davis, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Grady Memorial Hospital, Atlanta, Georgia
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Jacobi Medical Center, The Bronx, New York
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Houston Medical Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Point-of-care Ultrasound: Patient with suspected urolithiasis received ultrasonography performed in the emergency department.
  Ultrasonography in the Emergency Department: Perform ultrasonography in the ED (physician).
- Radiology Ultrasound: Patient with suspected urolithiasis received diagnostic ultrasonography in the radiology department.
  Diagnostic ultrasonography in radiology department: Diagnostic ultrasound completed in the radiology department at time 0.
- Computed Tomography: Patient with suspected urolithiasis received computed tomography in the radiology department.
  CT in Radiology: Computed tomography of abdomen completed in the radiology department at time 0.
Period: Overall Study
Arm/Group | Point-of-care Ultrasound | Radiology Ultrasound | Computed Tomography
Started | 909 | 901 | 966
Baseline Data Collection | 908 | 893 | 958
6-month Follow up | 876 | 843 | 923
Completed | 876 | 843 | 923
Not Completed | 33 | 58 | 43
Not completed — Lost to Follow-up | 17 | 36 | 21
Not completed — Withdrawal by Subject | 16 | 22 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Point-of-care Ultrasound | Radiology Ultrasound | Computed Tomography | Total
Number analyzed (Participants) | 908 | 893 | 958 | 2759
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (12.4) | 40.4 (12.8) | 40.7 (12.8) | 40.4 (12.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 12 | 21
  Between 18 and 65 years | 888 | 866 | 918 | 2672
  >=65 years | 16 | 22 | 28 | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 443 | 416 | 472 | 1331
  Male | 465 | 477 | 486 | 1428
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 8 | 18 | 38
  Asian | 35 | 39 | 51 | 125
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 4 | 6
  Black or African American | 236 | 213 | 241 | 690
  White | 587 | 593 | 616 | 1796
  More than one race | 32 | 33 | 23 | 88
  Unknown or Not Reported | 5 | 6 | 5 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 218 | 224 | 226 | 668
  Not Hispanic or Latino | 685 | 663 | 727 | 2075
  Unknown or Not Reported | 5 | 6 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 908 | 893 | 958 | 2759
History of Kidney Stones or Cancer [Number; unit: number of participants]
  Prior Kidney Stones | 377 | 385 | 387 | 1149
  No Kidney Stone | 531 | 508 | 571 | 1610
Self-Reported Pain Score [Mean (Standard Deviation); unit: units on a scale] — Range 0-10, higher numbers indicate more severe pain
  units on a scale | 8.3 (2.0) | 8.0 (2.4) | 8.1 (2.2) | 8.1 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: High Risk Diagnosis With Complication
Description: Missed or delayed diagnosis of appendicitis, pneumonia with sepsis, diverticulitis, abdominal aortic aneurysm with rupture, mesenteric ischemia with bowel perforation, renal infarction, stone with renal abscess, urosepsis/pyelonephritis with bacteremia, ovarian torsion with necrosis related to randomization and due to imaging modality.
Time Frame: 30 days from baseline
Measure: Number; unit: participants
Groups:
- Point-of-care Ultrasound: Patient with suspected urolithiasis will receive ultrasonography performed in the emergency department.
  Ultrasonography in the Emergency Department: Perform ultrasonography in the ED (physician).
Arm/Group | Point-of-care Ultrasound | Radiology Ultrasound | Computed Tomography
Number analyzed (Participants) | 908 | 893 | 958
participants | 6 | 3 | 2

2. Primary Outcome: Cumulative Radiation Exposure
Time Frame: Baseline plus 6 months post-baseline
Measure: Mean (Standard Deviation); unit: mSv
Arm/Group | Point-of-care Ultrasound | Radiology Ultrasound | Computed Tomography
Number analyzed (Participants) | 908 | 893 | 958
mSv | 10.1 (14.1) | 9.3 (13.4) | 17.2 (13.4)

3. Secondary Outcome: ED Length of Stay
Time Frame: Baseline visit excluding hospitalization
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Point-of-care Ultrasound | Radiology Ultrasound | Computed Tomography
Number analyzed (Participants) | 908 | 893 | 958
Hours | 5.1 [3.3 to 6.9] | 6.4 [4.6 to 8.2] | 6.3 [4.3 to 8.3]

4. Secondary Outcome: Return Visits to ED or Hospital
Time Frame: 6 months post-baseline
Measure: Number; unit: Number of visits
Arm/Group | Point-of-care Ultrasound | Radiology Ultrasound | Computed Tomography
Number analyzed (Participants) | 908 | 893 | 958
Number of visits
  Number of return visits to ED | 231 | 231 | 255
  Number of hospital readmissions | 87 | 84 | 83

5. Secondary Outcome: Accuracy for Stones by Arm
Time Frame: Up to 6 month follow-up for stone passage
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Point-of-care Ultrasound | Radiology Ultrasound | Computed Tomography
Number analyzed (Participants) | 908 | 893 | 958
Percent probability
  Sensitivity | 85 [80 to 89] | 84 [79 to 89] | 86 [82 to 90]
  Specificity | 50 [45 to 54] | 53 [49 to 57] | 53 [49 to 58]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Point-of-care Ultrasound | Radiology Ultrasound | Computed Tomography
Serious Adverse Events (participants affected / at risk) | 3/908 | 4/893 | 5/958
Other Adverse Events (participants affected / at risk) | 110/908 | 92/893 | 101/958
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Point-of-care Ultrasound (N=908) | Radiology Ultrasound (N=893) | Computed Tomography (N=958)
Acute Cholecystitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Renal Insuff/ Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian Torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Point-of-care Ultrasound (N=908) | Radiology Ultrasound (N=893) | Computed Tomography (N=958)
Unrelated Urosepsis Pyelonephritis (Renal and urinary disorders) | 5 (6) | 6 (8) | 4 (9)
Other - Various Unrelated (Renal and urinary disorders) | 105 (168) | 86 (117) | 97 (146) — Other various unrelated adverse effects, not categorized during study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No